CLINICAL TRIAL: NCT05576961
Title: Safety and Efficacy of Bacterial Strain RX-af01 Combined With PD-1 Antibody in Patients With Refractory Advanced Solid Tumors
Brief Title: Safety and Efficacy of RX-af01 Combined With PD-1 Antibody
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RX-af01-SYSUCC
Record Dates: First submitted 2022-09-16; First posted 2022-10-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor; Immune Checkpoint Inhibitor; Intestinal Flora
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: RX-af01 and toripalimab
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- regular dose of RX-af01 (Experimental): RX-af01 in combination with toripalimab
  Interventions: Drug: RX-af01
- high dose of RX-af01 (Experimental): 5 times dose of RX-af01 in combination with toripalimab
  Interventions: Drug: High dose RX-af01
- Mixed bacteria (Experimental): Mixed bacteria in combination with toripalimab
  Interventions: Drug: Mixed bacteria

INTERVENTIONS:
Drug: RX-af01 — Pretreatment： vancomycin: 125mg po, tid, D-6 to D-3 RX-af01: 2 capsules, bid, po, D-2 to D0 Treatment (Every 3 weeks) RX-af01: 1 capsule, bid, po, every day Toripalimab: 240mg, ivdrip, D1, every 3 weeks.
  Other Names: Toripalimab
  Arms: regular dose of RX-af01
Drug: Mixed bacteria — Pretreatment： vancomycin: 125mg po, tid, D-5 to D-3
  Other Names: Toripalimab
  Arms: Mixed bacteria
Drug: High dose RX-af01 — Pretreatment： vancomycin: 125mg po, tid, D-5 to D-3
  Other Names: Toripalimab
  Arms: high dose of RX-af01

SUMMARY:
This phase I trial evaluates the effects of RX-af01 in combination with toripalimab (PD-1 antibody), in treating patients with refractory advanced solid tumors, including melanoma, nasopharyngeal squamous carcinoma, esophageal squamous cell carcinoma, gastric adenocarcinoma, renal cell carcinoma, et al. RX-af01 is a kind of anti-tumor intestinal bacteria developed by our research group. Its main components are symbiotic bacteria from human intestine - Alisipes finegoldii (A. finegoldii.), which is a Gram negative anaerobic bacteria. Our previous research shows that A finegoldii. can significantly enhance the anti-tumor activity of PD-1 antibody in multiple mouse tumor models. Mechanism research shows that A finegoldii. can increase the infiltration of CD4 and CD8 positive immune cells in the tumor microenvironment, and enhances the anti-tumor activity of immune cells. The primary aim of this study is to explore the efficacy and safety of RX-af01 combined with PD-1 antibody in refractory advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase Ib study to evaluate the effects of RX-af01 in combination with toripalimab (PD-1 antibody), in treating patients with refractory advanced solid tumors, including melanoma, nasopharyngeal squamous carcinoma, esophageal squamous cell carcinoma, gastric adenocarcinoma, renal cell carcinoma, et al. This study will include 3 chorts. Cohort 1 uses the regular dose of RX-af01. Cohort 2 uses a high dose of RX-af01 which is 5 times of the regular dose of RX-af01. Cohort 3 uses a mixed bacteria including RX-af01, Bifidobacterium longum RX02 and Ligilactobacillus salivarius RX02.

Primary endpoint:

To determine the safety and efficacy of bacterial strain RX-af01 in combination with toripalimab in refractory advanced solid tumors.

Secondary endpoint:

1. Progression free survival (PFS)
2. Overall survival (OS)
3. Duration of response (DOR)
4. Tumor microenvironment
5. Changes in flora species/abundance

ELIGIBILITY:
Inclusion Criteria:

* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] stage IV) solid tumors, including melanoma, nasopharyngeal squamous carcinoma, esophageal squamous cell carcinoma, gastric adenocarcinoma, renal cell carcinoma, et al.
* Fail to or could not tolerate standard treatment.
* Receive at least 2 cycles of PD-1/PD-L1/CTLA4 inhibitors and the response is complete response (CR) or partial response (PR) or stable disease (SD).
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Recovery to baseline or =< grade 1 CTCAE v5 from toxicities related to any prior treatments unless adverse events (AE[s]) are clinically nonsignificant and/or stable on supportive therapy
* ECOG performance status score: 0-1
* Males and females, ages >= 18
* Absolute neutrophil count (ANC) >= 1500/uL without granulocyte colony-stimulating factor support (within 14 days before first dose of study treatment)
* Platelets >= 90,000/uL without transfusion (within 14 days before first dose of study treatment)
* Hemoglobin >= 8 g/dL (>= 80 g/L) (within 14 days before first dose of study treatment)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) =< 3 x upper limit of normal (ULN). ALP =< 5 x ULN with documented bone metastases (within 14 days before first dose of study treatment) Total bilirubin =< 1.5 x ULN (for subjects with Gilbert's disease =< 3 x ULN) (within 14 days before first dose of study treatment)
* Serum albumin >= 3.0 g/dl (within 14 days before first dose of study treatment)
* Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN (within 14 days before first dose of study treatment)
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance >= 40mL/min (>= 0.675 mL/sec) using the Cockcroft-Gault equation (within 14 days before first dose of study treatment)
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg (=< 113.2 mg/mmol), or 24-hour (h) urine protein =< 1 g (within 14 days before first dose of study treatment)
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of treatment, 5 months after the last dose of PD-1 inhibitor for women with childbearing potential, and 7 months after the last dose of PD-1 inhibitor for men
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating [FSH] level > 40 mIU/mL to confirm menopause).

Exclusion Criteria:

* Current use, or intent to use, probiotics, yogurt, or bacterial fortified foods during the period of treatment
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  1. Cardiovascular disorders:

     Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.
  2. Subjects with a diagnosis of incidental, subsegmental pulmonary embolism (PE) or deep vein thrombosis (DVT) within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation for at least 1 week before first dose of study treatment.
  3. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment

* Other clinically significant disorders that would preclude safe study participation:

Any active, known, or suspected autoimmune disease will be excluded, with the following exceptions: Type 1 diabetes mellitus; hypothyroidism only requiring hormone replacement; skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment; conditions not expected to recur in the absence of an external trigger.

* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before first dose of study treatment. Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed.
* Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection (with the DNA copy number >1000 copies/ml), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection.
* Serious non-healing wound/ulcer/bone fracture.
* Malabsorption syndrome.
* Uncompensated/symptomatic hypothyroidism.
* Moderate to severe hepatic impairment (Child-Pugh B or C).
* Requirement for hemodialysis or peritoneal dialysis.
* History of solid organ or allogenic stem cell transplant.
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal, or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment. Furthermore, subjects with a history of additional risk factors for torsades de pointes (e.g., long QT syndrome) are also excluded.
* Pregnant or lactating females
* Inability to swallow tablets or unwillingness or inability to receive IV administration
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies.
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 5 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 1 year
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, including complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 1 year
  From the time of enrollment to the date of death or last followup.
Progression free survival (PFS) | Up to 1 year
  From the time of enrollment to the date of disease progression or death or last followup.
Duration of response (DoR) | Up to 1 year
  The time from the first assessment of CR or PR to the first assessment of PD or death (caused by any reason)
Change of tumor microenvironment | Up to 1 year
  Infiltration of immune cells, including CD8+T cell, Treg cell et al.
Comparison of the Shannon index (a measure of microbial diversity) | Up to 1 year
  Using translational methods, will compute the Shannon index at baseline for a comparison of microbial diversity.

CONTACTS AND LOCATIONS:
Locations (1):
- Miao-Zhen Qiu, Guangzhou, Guangdong, China